CLINICAL TRIAL: NCT01090934
Title: Etude de la Performance Diagnostique de l'EEG-Haute Résolution Sur la Localisation de la Zone épileptogène Pour le Traitement Chirurgical Des épilepsies Partielles Pharmaco-résistantes
Brief Title: Localizing the Epileptogenic Zone With High Resolution Electroencephalography
Acronym: EEG-HR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University Hospital, Marseille (Other); CHU de Reims (Other); Centre National de la Recherche Scientifique, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, louis maillard, Dr Louis MAILLARD, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-A00574-53
Record Dates: First submitted 2010-02-05; First posted 2010-03-23 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Partial Epilepsy
Keywords: Diagnosis; Partial Epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high resolution EEG (Experimental)
  Interventions: Device: High Resolution EEG
- Stereo Electroencephalography (Active Comparator)
  Interventions: Device: Stereo-electroencephalography

INTERVENTIONS:
Device: High Resolution EEG — High Resolution EEG
  Other Names: electrical source imaging
  Arms: high resolution EEG
Device: Stereo-electroencephalography — SEEG
  Other Names: depth-electroencephalography
  Arms: Stereo Electroencephalography

SUMMARY:
Multicenter prospective study comparing the diagnosis value of high-resolution EEG and depth-EEG to localize the epileptogenic zone in drug resistant partial epilepsies.

ELIGIBILITY:
Inclusion Criteria:

* medically intractable patial epilepsy confirmed by video-EEG recordings of epileptic seizures.
* Depth EEG (Stereo-EEG) required to delineate the epileptogenic zone and define the surgical procedure.
* full informed consent of the patient (or of his/ her legal representative)
* 15 year or older patient

Exclusion Criteria:

* contraindication to cortectomy
* contraindication to depth-EEG
* indication of epilepsy surgery without depth-EEG monitoring
* high grade glioma, arterio-veinous malformations

  * pregnancy
  * history of severe cardio-vascular event (coronaropathy, stroke)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-10; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of electrical source localization of inter-ictal and ictal discharges using high-Resolution EEG for localizing the epileptogenic zone (the stereo-electroencephalography will be the reference method) | 3 years
  results of electrical sources localization of inter-ictal and ictal discharges are compared to the epileptogenic zone defined by SEEG

SECONDARY OUTCOMES:
inter-observer reliability of electrical source localization of inter-ictal and ictal discharges for localizing the epileptogenic zone. | 3 years
  sources localization of inter-ictal and ictal discharges will be interpreted by two independant epileptologists, blinded to the results of stereo-EEG.
sensitivity and specificity of high resolution EEG and electrical source imaging for surgical decision | 3 years
  decision of surgery and the limits of the cortectomy established with electrical source imaging will be compared to the decision of surgery and the limits of the cortectomy established with Stereo-electroencephalography.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Maillard, MD, PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (2):
- France (2):
  - University Hospital of Marseille, Marseille
  - Central Hospital, Nancy

REFERENCES:
- [Background] Maillard L, Koessler L, Colnat-Coulbois S, Vignal JP, Louis-Dorr V, Marie PY, Vespignani H. Combined SEEG and source localisation study of temporal lobe schizencephaly and polymicrogyria. Clin Neurophysiol. 2009 Sep;120(9):1628-36. doi: 10.1016/j.clinph.2009.06.022. Epub 2009 Jul 24. PMID 19632148
- [Background] Koessler L, Benar C, Maillard L, Badier JM, Vignal JP, Bartolomei F, Chauvel P, Gavaret M. Source localization of ictal epileptic activity investigated by high resolution EEG and validated by SEEG. Neuroimage. 2010 Jun;51(2):642-53. doi: 10.1016/j.neuroimage.2010.02.067. Epub 2010 Mar 4. PMID 20206700
- [Result] Koessler L, Cecchin T, Caspary O, Benhadid A, Vespignani H, Maillard L. EEG-MRI co-registration and sensor labeling using a 3D laser scanner. Ann Biomed Eng. 2011 Mar;39(3):983-95. doi: 10.1007/s10439-010-0230-0. Epub 2010 Dec 8. PMID 21140291
- [Result] Koessler L, Salido-Ruiz R, Ranta R, Louis-Dorr V, Gavaret M, Maillard L. Influence of source separation and montage on ictal source localization. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:2898-901. doi: 10.1109/IEMBS.2010.5626321. PMID 21095980